CLINICAL TRIAL: NCT05808985
Title: Intestinal Microbiome-based Research for the Prevention of Acute Graft-versus-host Disease
Brief Title: Intestinal Microbiome-based Research for the Prevention of Acute GVHD
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Soonchunhyang University Hospital (Other)
Responsible Party: Principal Investigator, Seug yun Yoon, MD, assistant professor, Soonchunhyang University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2022-06-011
Record Dates: First submitted 2023-01-27; First posted 2023-04-12 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-01

CONDITIONS: Graft Versus Host Disease; Postbiotics; Butyrate
Keywords: butyrate; Graft Versus Host Disease; postbiotics
MeSH Terms: conditions — Graft vs Host Disease | interventions — Butyric Acid

STUDY DESIGN:
Intervention Model Description: Take butyric acid (sodium butylate 600mg 2 tablets, BodyBio⒭)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Butyrate (Experimental): Take butyric acid (sodium butylate 600mg 2 tablets, BodyBio⒭ per day)
  Interventions: Drug: sodium butyrate

INTERVENTIONS:
Drug: sodium butyrate — Take butyric acid (sodium butylate 600mg 2 tablets, BodyBio⒭, per day)

SUMMARY:
Hematopoietic stem cell transplantation consists of preconditioning chemotherapy, stem cell infusion, and engraftment of hematopoietic stem cells. In this process, in the case of recipients who receive hematopoietic stem cells, their immune system is completely destroyed and then undergoes a situation in which it is reconstituted. In this process, the diversity of the intestinal microbiome is reduced, and it is widely known that a severe decrease is associated with the occurrence of an acute graft-versus-host reaction. Attempts to improve the intestinal microbiome include prebiotics, probiotics, and postbiotics. Prebiotics can be expected to improve the intestinal microbiome by acting as nutrients for beneficial bacteria in the intestine, but their role may be limited in situations where the diversity of the intestinal microbiome has already decreased. Probiotics are a method to expect improvement of the intestinal microbiome by administering the beneficial bacteria themselves in the intestine, but there is a difficulty in reaching the intestine properly through stomach acid, and there is a risk of causing sepsis in immunocompromised patients. Postbiotics is a product that beneficial bacteria metabolize and release prebiotics in the intestine, and the microbiome in the intestine is actually responsible for the function that affects the human body. Therefore, in this study, postbiotics are administered to patients undergoing hematopoietic stem cell transplantation who are concerned that the diversity of the intestinal microbiome may have already decreased, to improve the intestinal microbiome and hope to prevent graft-versus-host reactions through this. Furthermore, it is intended to improve the outcome of allogeneic hematopoietic stem cell transplantation.

DETAILED DESCRIPTION:
1. step After explaining the background and purpose of the study to the subjects undergoing hematopoietic stem cell transplantation at Soonchunhyang University Seoul Hospital and obtaining consent, before transplantation (D-7), on the day of transplantation (D0), and at the time of engraftment after transplantation (D+ 14), 30 days after transplantation (D+30), 3 months after transplantation (D+90), if complications occur after a total of 5 times, if the researcher deems it necessary, with the consent of the patient, additional feces are collected. About 10g per dose will be received and stored in a freezer at the Institute of Clinical Molecular Biology, Soonchunhyang University until December 2027, and DNA will be extracted and microbiome analyzed later, and discarded at the end of the study. In the process of allogeneic hematopoietic stem cell transplantation, the subjects had difficulty in oral intake during the transplantation process after pretreatment chemotherapy, so at the time of engraftment oral intake was possible, starting to take butyric acid (sodium butylate 600mg 2 tablets, BodyBio⒭) for 3 months after transplantation Continue taking until All expenses incurred in the course of testing are borne by the researcher. The patient's clinical progress and test results related to hematopoietic stem cell transplantation are investigated based on medical records.
2. Duration of subject participation and expected number of subjects For patients undergoing hematopoietic stem cell transplantation at our hospital from the date of IRB approval to December 2023 (About 20 patients a year receive hematopoietic stem cell transplantation at our center, and it is expected that about 30 patients will participate)
3. Clinical Study Restrictions and Subject Obligations Subjects who agreed to the study must take butyric acid (sodium butylate 600mg 2 tablets, BodyBio⒭) from the time of engraftment to 3 months after transplantation, and must collect and submit feces at the designated time and in an appropriate way.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing hematopoietic stem cell transplantation
* Adult patients over 19 years and under 70 of age

Exclusion Criteria:

* Patients who did not agree to participate in the study
* If feces are not suitable for analysis

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2022-09-02 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of GVHD | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Jong-Ho Won, MD, PhD, Study Chair — Soonchunhyang University Hospital
Locations (1):
- Soonchunhyang University Seoul Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No